CLINICAL TRIAL: NCT01073098
Title: Evaluation of Muscle StO2 as a Prognostic Factor After Out of Hospital Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Clinical Research and Innovation (Other)
Collaborators: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor-Investigator, Department of Clinical Research and Innovation, Department of Clinical Research and innovation (drc), Centre Hospitalier Universitaire de Nice
Organization: Centre Hospitalier Universitaire de Nice (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2009-A01187-50
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2011-12

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Vascular occlusion test — Reperfusion slope after vascular occlusion test

SUMMARY:
Out of hospital cardiac arrest is a major health problem. Prognosis is still poor even after return to spontaneous circulation. The pathophysiology of cardiac arrest implies ischemia-reperfusion and sepsis like syndrome. These phenomenons can lead to microvascular dysfunction explaining probably multi-organ failure after cardiac arrest. Few means allow the exploration of microvascular function in human. Muscle StO2 is a technique allowing the assessment of microvascular function non-invasively. The aim of this study is to evaluate muscle StO2 as a prognostic factor after out of hospital cardiac arrest.

DETAILED DESCRIPTION:
Out of hospital cardiac arrest is a major health problem accounting for 375000 deaths each year in Europe. Even after return to spontaneous circulation, survival is poor because of complications such as post-anoxic encephalopathy and multi-organ failure. The pathophysiology of cardiac arrest implies ischemia-reperfusion and sepsis like syndrome. These conditions are frequently associated with microvascular dysfunction that can be the "motor" of multi-organ failure. Few means allow the exploration of microvascular function in human. Recently, StO2, a non-invasive technique assessing microvascular function has been described. This technique measures the tissular saturation of a muscle using the near-infrared spectroscopy technique. It has been described to be a good prognostic factor during haemorrhagic shock state. Dynamic parameters such as reperfusion slope allow discriminating between survivors and survivors after severe sepsis. This dynamic test assesses the microvasculature recruitment that could be a marker of better prognosis. The aim of this study is to evaluate muscle StO2 as a prognostic factor after out of hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Out of hospital cardiac arrest
* Patient aged between 18 and 80 years
* Having a Social Security System

Exclusion Criteria:

* Pregnant women, lack of appropriate consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Reperfusion slope after vascular occlusion test. This parameter will be compared between survivors and non-survivors | Four measurements : on admission, since the body core temperature reaches 34°, after 24 hours of hypothermia and 48 hours after admission to ICU

SECONDARY OUTCOMES:
Muscle StO2 during the first 2 days Lactatemia during the first 2 days These parameters will be compared between survivors and non-survivors | Muscle StO2 will be monitored continuously during the first 2 days Lactatemia will be measured every 12 hours until normalization

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe ORBAN, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - CHU de Nice -Hôpital l'Archet, Nice
  - CHU de Nice Hôpital Saint Roch, Nice